CLINICAL TRIAL: NCT03577873
Title: Randomized Controlled Trial on Necessity of Cholecystectomy for Patients With Bile Duct Stones Combined With Gallbladder Stones After Clearance of Stones
Brief Title: RCT on Necessity of Cholecystectomy for Patients After Clearance of Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Deputy director, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-107-01
Record Dates: First submitted 2018-06-05; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Gallbladder Stones; Complication; Cholecystectomy
Keywords: gallbladder stones; common bile duct stones; Endoscopic retrograde cholangiopancreatography
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gallbladder preserved (Placebo Comparator): Patients with stones in their bile ducts and gallbladders will keep gallbladders in stay after clearance of bile duct stones with ERCP.
  Interventions: Other: gallbladder preserved
- cholecystectomy (Experimental): Patients with stones in their bile ducts and gallbladders will undergo cholecystectomy after clearance of bile duct stones with ERCP.
  Interventions: Procedure: cholecystectomy

INTERVENTIONS:
Other: gallbladder preserved — Gallbladders will be remained after clearance of bile duct stones with ERCP and conventional therapy, such as fluid replacement and prophylactic anti infection, will be accepted.
  Arms: gallbladder preserved
Procedure: cholecystectomy — Cholecystectomy will be done right now after clearance of bile duct stones with ERCP, and then conventional therapy will be accepted.
  Arms: cholecystectomy

SUMMARY:
To discuss necessity of cholecystectomy for patients with stones in their bile ducts and gallbladders in the absence of absolute operation indications of cholecystectomy after clearance of bile duct stones with ERCP.

DETAILED DESCRIPTION:
Cholecystectomy was recommended for patients with stones in their bile ducts and gallbladders in European and American countries after clearance of bile duct stones with ERCP, which reduced the incidence of biliary events. However, some researches showed that the incidence of biliary events was not reduced but increased.The purpose of this study is to discuss the necessity of cholecystectomy for patients with stones in their bile ducts and gallbladders in the absence of absolute operation indications of cholecystectomy after clearance of bile duct stones with ERCP.

ELIGIBILITY:
Inclusion Criteria:

Obtention of a written informed consent; Clinical diagnosis of gallbladder stones and common bile duct stones; No absolute operation indications of cholecystectomy

Exclusion Criteria:

Intrahepatic stones; Malignant tumor disease ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
biliary events | 12 months
  The incidence of biliary events will be compared in the two groups.

SECONDARY OUTCOMES:
adverse events | 12 months
  Number of participants with adverse events: type, frequency and intensity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangfeng Zhang, M.S, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heo J, Jung MK, Cho CM. Should prophylactic cholecystectomy be performed in patients with concomitant gallstones after endoscopic sphincterotomy for bile duct stones? Surg Endosc. 2015 Jun;29(6):1574-9. doi: 10.1007/s00464-014-3844-8. Epub 2014 Oct 8. PMID 25294531